CLINICAL TRIAL: NCT06172803
Title: RESToRE: Restoring Energy With Sub-symptom Threshold Optimized Rehabilitation Exercise for Long COVID
Brief Title: Restoring Energy With Sub-symptom Threshold Optimized Rehabilitation Exercise for Long COVID
Acronym: RESToRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAU4504 (Aim 1)
Record Dates: First submitted 2023-12-14; First posted 2023-12-15 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Long Covid19; Exercise Intolerance; Riboflavin-Responsive
Keywords: Riboflavin; Rehabiliation; Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Restore polishing paste; Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RESToRE (Experimental): Participants will receive RESToRE, an interdisciplinary, hybrid 8- week intervention.
  Interventions: Behavioral: Restoring Energy with Sub-symptom Threshold Aerobic Rehabilitation Exercise
- Light Stretching Exercise (Active Comparator): The control group will receive 8-week, attention-matched, stretching and breathing exercises, supervised by a rehabilitation clinician.
  Interventions: Behavioral: Light Stretching/Breathing Exercises

INTERVENTIONS:
Behavioral: Restoring Energy with Sub-symptom Threshold Aerobic Rehabilitation Exercise — 8 week exercise program. 20 minutes of home aerobic exercise most days, phone- based motivational exercise coaching and supervised exercise with our team exercise physiologist.
  Other Names: RESToRE
  Arms: RESToRE
Behavioral: Light Stretching/Breathing Exercises — The control group will receive 8-week, attention-matched, stretching and breathing exercises, supervised by a rehabilitation clinician (via 20-minute weekly video visits). Exercises performed 5 days a week will not increase HR significantly. Participants will record and track their HR with Apple watch and app; like RESToRE, fidelity of treatment will be objectively measured using HR data.
  Arms: Light Stretching Exercise

SUMMARY:
The overall goal of this study is to find out if rehabilitation exercise can help people who have long COVID. Participants will be randomized by chance to receive either aerobic exercise or breathing exercise (combined with stretches). Participants will be guided and supported in completing a tailored, 6-week home exercise program to be performed 5 - 6 days a week, prescribed and supervised by rehabilitation therapists. Participants will perform breathing exercises, which will be supervised by an occupational therapist. The focus of Aim 1 is to determine feasibility of implementing RESToRE in long COVID.

DETAILED DESCRIPTION:
Long COVID, also known as post-acute coronavirus 2019 syndrome, is characterized by debilitating, multi-organ symptoms beyond 3 months from the onset of acute illness, consistent with autonomic nervous system dysfunction. Prevalence estimate of long COVID is 10 - 20% of survivors of COVID-19, representing about 10-20 million global long-term cases. Multi-organ, autonomic-related symptoms of long COVID, such as exhausting fatigue and post-exertional malaise, are remarkably like post-concussion syndrome and chronic fatigue syndrome. Post-exertional malaise, likely a cardinal symptom of long COVID, is "an exacerbation of some or all of an individual's symptoms after physical or cognitive exertion, or orthostatic stress", significantly impacting functional ability and quality of life. This abnormal response to exertion is often described as "flu-like" and typically includes brain fog. Common "long hauler" symptoms reported in our cohort of patients with long COVID (n=30) were fatigue (>70%), symptoms of dysautonomia (80%, primarily orthostasis), "brain fog" (100%), and new or worse mood symptoms (90%), especially anxiety. Experience from Severe Acute Respiratory Syndrome (SARS-CoV-1) notably showed that survivors suffered chronic fatigue and mental illnesses 4 years after acute viral illness. Rehabilitation studies in coronavirus disease (Covid-19) have targeted sub-acute lung sequelae of Covid-19 rather than post-acute sequalae of long COVID. This study addresses the World Health Organization's urgent call for rehabilitation research for long COVID.

The investigators identified blunted rise in heart rate (HR), called chronotropic intolerance, during maximal cardiopulmonary exercise testing (CPET) in 19 adults with long COVID. Chronotropic intolerance is defined as inability to meet 80% of age-derived heart rate, HR peak. Group HR peak mean (SD) was 69 (7.7) % predicted. This blunted rise in HR is associated with post-exertional malaise, similar to the pattern of symptoms in post-concussion syndrome and chronic fatigue syndrome, which share underlying autonomic nervous system (ANS) dysfunction and impaired cerebral blood flow regulation. The investigators identified a need for more comprehensive and precise measurement of post-exertional malaise in long COVID. In a randomized controlled trial (RCT), the investigators also tested a sub-symptom threshold aerobic exercise program, focused on treating persisting symptoms of post-concussion syndrome. The investigators found this aerobic exercise program reduced persistent symptoms of exercise intolerance, fatigue, and dysautonomia more quickly in subjects compared with a control group of stretching exercises (n=103).

Informed by research in post-concussion syndrome, the investigators are proposing a two-arm randomized controlled trial (RCT) to study the feasibility of an exercise program called, Restoring Energy with Sub-symptom Threshold Aerobic Rehabilitation Exercise (RESToRE). The central hypothesis is that restoration of autonomic control through RESToRE will resolve persisting symptoms of long COVID faster compared with placebo-like stretching and breathing exercise (without rise in HR). RESToRE is an interdisciplinary, hybrid 8-week intervention consisting of three core components: (1) home-based aerobic exercise, of 20 minutes most days, with HR monitoring at 70-80% of the HR threshold at which symptoms increase, (2) phone-based motivational exercise coaching, 20 minutes weekly; and (3) supervised exercise with an exercise physiologist, twice-monthly in the clinic. Key to RESToRE's feasibility is its telehealth component, including Apple watch and app for HR fidelity monitoring, PhysiTrack's exercise library app, and LifeData dashboard for real-time post-exertional malaise and remote exercise monitoring. Our long-term goal is to establish an efficacious exercise program to speed recovery from long COVID.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Age of 21 years or older
* Diagnosis of long COVID
* Score >0 on energy, daily activities, sleep, chest tightness, or breathlessness on COPD Assessment Test or self-reported brain fog
* Able to use a smartphone.

Exclusion Criteria:

* >70years old due to risk of sarcopenia
* Frailty defined as gait speed <1 m/s on 4- Meter Gait Speed (4MGS) test due to falls risk
* Diagnosis of chronic cardiac or pulmonary disease, including atrial fibrillation, ME/CFS, post-concussion syndrome, chronic Lyme disease, lupus, or sarcopenia comorbidities (due to PEM and/or fatigue)
* Medical history of ICU stay for COVID-19 illness due to risk of post-ICU syndrome and increased rehabilitation needs
* Inability to ambulate independently and safely without a walking aide
* Diagnosis of dementia or neurodegenerative disease, multiple sclerosis, or rheumatoid arthritis with associated cognitive dysfunction or fatigue.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Number of participants who enrolled | 10 weeks
  Feasibility of the RESToRE program will be determined by measuring the number of participants who enroll.
Number of participants who completed | 10 weeks
  Feasibility of the RESToRE program will be determined by measuring the number of participants who complete (participated through the end of the study).
Number of participants who adhered to session attendance | 10 weeks
  Feasibility of the RESToRE program will be determined by measuring the number of participants who achieve ≥80% exercise adherence and session attendance.

SECONDARY OUTCOMES:
PROMIS-29 scale score | baseline and post intervention at 8 weeks
  This toll/questionnaire is designed to measure participants quality of life. Score range is 1-5, with higher score correlating to worse outcomes.
Rand 36-Item Health Survey (SF-36) score | Baseline and Post Intervention at 8 weeks
  This survey evaluates participants mental and physical health with 8 scales aggregated. Score range is 1-6, with the higher score correlating to worse overall health outcomes.
VO2 % predicted from Cardiopulmonary Exercise Testing (CPET) | Baseline and post intervention at 8 weeks
  VO2 % predicted (oxygen consumption) based on normative data. Participants' scores will be compared to norms for assessing exercise ability. Group means will be compared.
Number of participants with orthostatic hypocapnia. | baseline and post intervention at 8 weeks
  The Nasa Lean Test: Participants will stand and lean against a wall with shoulder blades touching and heels 6 - 8 inches from the wall for 10 minutes. HR, BP, SpO2, ETCO2, and symptoms will be recorded in standing leaning posture every minute for 10 mins. Capnography will be used to identify orthostatic hypocapnia.
EuroQol: Education Quotient-5D Visual Analogue Scale score | baseline and post intervention at 8 weeks
  This is to measure quality of life. Score range is 0-100, with 100 being the best health you can imagine and 0 being the worst health.
General Symptom Questionnaire (SGQ-30) score | baseline and post intervention at 8 weeks
  This is to assess participants symptoms regarding pain/fatigue, psychiatric, neurological, and viral-like. Score range is 0 which is not at all to 4 which is very much. Higher score represents worst symptoms.
PROMIS Cognitive Function score | baseline and post intervention at 8 weeks
  This is an 8-item Short Form, measuring perceived difficulties in cognition (e.g., attention, concentration, executive functioning). Score range is 1-5. 1 is very often to 5 which is never. The higher score is better.
Global Change Assessment (GCA) score | baseline and post intervention at 8 weeks
  This is to measure patients change of symptoms in terms of physical function and fatigue throughout the study. Score range is -7 to 7. -7 is a very great deal worse and 7 is a great deal better. The higher the score the better.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Norweg, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States